CLINICAL TRIAL: NCT03484312
Title: Hypertensive Urgency Treatment and Outcomes in a Northeast Thai Population: The Results From the Hypertension Registry Program
Brief Title: Hypertensive Urgency Treatment and Outcomes in a Northeast Thai Population
Status: Completed | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Praew Kotruchin, Associate professor, Khon Kaen University
Other Study IDs: HE591508
Record Dates: First submitted 2018-03-15; First posted 2018-03-30 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Hypertension on Emergence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies have reported a high prevalence of hypertensive (HT) urgency. However, these studies have also reported low rates of serious complications, suggesting that rapid blood pressure (BP) reduction may be unnecessary. There are limited clinical data available on this topic in Asian populations. The investigators aimed to determine the basic characteristics, treatment methods, and outcomes in HT urgency patients, both in the emergency room (ER) and at a two-week follow-up.

DETAILED DESCRIPTION:
Previous studies have reported the high prevalence of hypertensive (HT) urgency. However, these studies have also reported low rates of serious complications, suggesting that rapid blood pressure (BP) reduction may be unnecessary. There are limited clinical data available on this topic in Asian populations. The investigators aimed to determine the basic characteristics, treatment methods, and outcomes in HT urgency patients, both in the emergency room (ER) and at a two-week follow-up.

This was a cohort study conducted at Srinagarind hospital, a tertiary-care level university hospital in Khon Kaen, Thailand. The data collection period was from January 2012 to June 2017. The Khon Kaen University Ethics Committee in Human Research approved the protocol. Patients aged 18 years or older who visited the ER with a diagnosis of HT urgency were consecutively enrolled in the study. Patients who were pregnant or lactating had secondary causes of HT, or had incomplete medical records were excluded from the study Office BP was measured using an upper arm cuff oscillometric BP device. The appropriate cuff size for each individual's arm circumference was used. Three BP readings were taken at 30-second intervals with the patient in a sitting position after five minutes of rest. The average of three BP measurements was used for analysis.

Baseline characteristic data were shown as the mean and standard deviation (SD) or percentage. An independent sample t-test was used to compare between groups for continuous variables including age, body mass index (BMI), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), time of treatment, and the number of medications being administered. A probability value <0.05 was considered statistically significant. All statistical analyses were performed with SPSS for Mac version 20.0, registered to Khon Kaen University.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older who visited the ER with a diagnosis of HT urgency

Exclusion Criteria:

* Pregnant or lactating
* Secondary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older who visited the ER with a diagnosis of HT urgency were consecutively enrolled in the study. Patients who were pregnant or lactating, had secondary causes of hypertension were excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure (mm Hg) | Up to 24 hours
  The investigators aimed to compare systolic and diastolic blood pressure level at baseline and before discharge from the emergency room (ER)
Discharge status including 1. discharge to home 2. admit to hospital 3. death 4. refer to another hospital | Up to 24 hours
  Discharge status from emergency room was observed and collected.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure at first hypertension clinic follow up | 2 weeks after discharge from emergency room
  Office systolic and diastolic blood pressure at first clinic follow up (2 weeks after emergency room visit)

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Medicine, Khon Kaen University, Khon Kaen, Muang, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Data will be provided upon a requested
Supporting Information: Study Protocol
Time Frame: 1 year